CLINICAL TRIAL: NCT07217080
Title: Thalamocortical Interactions and the Effect of Thalamic Stimulation on Sleep Oscillations
Brief Title: The Effect of Thalamic Stimulation on Sleep Oscillations
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rina Zelmann, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007P000165-1R01AG090302; 1R01AG090302 (NIH)
Record Dates: First submitted 2025-10-10; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Sleep; Neuromodulation
Keywords: Sleep; Spindles; Thalamus; electroencephalography; intracranial EEG; Neuromodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalamic stimulation to evoke or disrupt sleep spindles (Experimental): Stimulation of thalamic nuclei and cortical structures using electrical stimulation.
  Interventions: Behavioral: Effect of Electrical Stimulation on Sleep

INTERVENTIONS:
Behavioral: Effect of Electrical Stimulation on Sleep — Direct electrical stimulation of thalamic nuclei and cortical structures using clinically implanted depth electrodes will allow assessing the effect of stimulation on sleep oscillations.

SUMMARY:
The thalamus plays a key role in supporting sleep and is also a target of therapeutic stimulation. This project investigates when, where, and how electrical stimulation delivered to the thalamus in humans elicits or disrupts sleep oscillations. This research is a first step to better understand how current neuromodulation therapies affect sleep and may help advance toward new therapies to improve sleep for a wide range of neurological and neuropsychological disorders.

DETAILED DESCRIPTION:
The thalamus plays a key role in supporting sleep. The thalamus is also increasingly used as a stimulation therapeutic target, but the effect of thalamic stimulation on sleep has not been investigated.

We hypothesize that electrical stimulation delivered to the thalamus in humans could both elicit and disrupt sleep oscillations, such as spindles, depending on the timing and location of stimulation. We propose a study to obtain direct evidence in humans of how thalamic stimulation affects sleep.

We will test the hypothesis that stimulation during a thalamic sleep spindle disrupts it, while stimulation outside evokes a response resembling a k-complex followed by a spindle. Participants will be patients with refractory epilepsy who have semi-chronically implanted depth electrodes in the thalamus and other brain regions (~100) as part of the pre-surgical clinical work-up. We will detect spindles and stimulate during or outside oscillations using a real-time closed-loop system that we developed. Simultaneously recording across the brain will comprehensively map the effect and extent of thalamic stimulation on sleep oscillations.

This will be the first step to unravel the effect of thalamic stimulation on sleep oscillations and maintenance. This will increase our understanding of the thalamus as a relay of sleep oscillations and could have profound implications to ensure good sleep quality for the increasing number of people implanted with therapeutic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients getting intracranial recordings for clinical purposes who, as part of that plan, will receive thalamic electrodes.

Exclusion Criteria:

* previous extensive resection or large atrophy

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from pre-stimulation baseline of sleep spindle rate | 10 to 3000 milliseconds following stimulation
  An increase in spindle rate is achieved if at least 50% of trials evoke a spindle as measured on intracranial EEG following stimulation. A spindle is evoked when the power in the 10-16Hz band is larger than pre-stimulation baseline power by at least 2 standard deviations.

SECONDARY OUTCOMES:
Number of channels with responses to stimulation | 10 to 3000 milliseconds following stimulation
  A channel responds to stimulation if the broadband power is larger than baseline by at least 2 standard deviations, as measured from the intracranial EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Zelmann, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-identified intracranial EEG recordings will be collated across participants. Data used in the results publication will be shared.
Supporting Information: Analytic Code
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: We will share electrophysiological data with the scientific community via the Data Archive for the BRAIN Initiative (DABI), or another NIH-approved database, where we will offer access to our database of neural activity.